CLINICAL TRIAL: NCT06790498
Title: A Long-Term Follow-up Study of Participants Exposed to Renal Autologous Cell Therapy From Studies REGEN-006, REGEN-007, and REGEN-015 (REGEN-008S2)
Brief Title: Long-Term Follow-up Study of Participants Exposed to Renal Autologous Cell Therapy Frozen Product
Status: Enrolling by invitation | Type: Observational
Sponsor: Prokidney (Industry)
Responsible Party: Sponsor
Other Study IDs: REGEN-008S2
Record Dates: First submitted 2025-01-14; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Diabetic Kidney Disease; Chronic Kidney Disease
MeSH Terms: conditions — Diabetic Nephropathies; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Research samples (serum/plasma and/or urine) will be collected, frozen, and stored for the future research. Participating participants can opt out of long-term storage of their unused specimens during the informed consent process or at any time during the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CKD patients previously treated with REACT: Participants Exposed to Renal Autologous Cell Therapy from studies REGEN-007, REGEN-006, REGEN-015 (REGEN-008S2).
  Interventions: Biological: Renal Autologous Cell Therapy (REACT)

INTERVENTIONS:
Biological: Renal Autologous Cell Therapy (REACT) — No interventions in this trial

SUMMARY:
The purpose of this study is to evaluate the long-term safety, efficacy, and durability in participants with chronic kidney disease (CKD) who received up to four REACT injections, delivered percutaneously into either the same or bilateral kidneys in previous studies.

DETAILED DESCRIPTION:
This observational extension study is a multi-center, prospective, non-therapeutic study, where up to 50 participants who have been enrolled and dosed with Renal Autologous Cell Therapy in previous interventional clinical studies (REGEN-007, REGEN-006, REGEN-015) will be monitored for up to five years with alternating in clinic and phone visits.

ELIGIBILITY:
Inclusion Criteria:

* The participant must have received REACT in a previous trial (REGEN-006, REGEN- 007, and REGEN-015) for the treatment of chronic kidney disease and completed an end of study visit in their previous trial per protocol.
* The participant is willing and able to cooperate with all aspects of the protocol.
* The participant is willing and able to provide signed informed consent.

Exclusion Criteria:

• Participant did not receive REACT in a previous trial for the treatment of chronic kidney disease

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Chronic Kidney Disease
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2030-05-31 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
Long-term safety of REACT follow-up after completing their enrollment in the investigational clinical studies. | 60 months from completion of parent protocol EOS Visit
  Evaluation of the long-term safety of REACT will be assessed via:
  * Incidence of delayed serious adverse events (SAEs) obtained throughout long-term follow-up after completing their enrollment in the investigational clinical studies.
  * Incidence of delayed biopsy-related SAEs obtained throughout long-term follow-up after completing their enrollment in the investigational clinical studies.
  * Incidence of delayed injection procedure related SAEs obtained throughout long-term follow-up after completing their enrollment in the investigational clinical studies.
  * Incidence of delayed investigational product related SAEs obtained throughout long-term follow-up after completing their enrollment in the investigational clinical studies.

SECONDARY OUTCOMES:
Time from first injection to eGFR <15 mL/min/1.73m² using the 2009 CKD-EPI serum creatinine equation. | 60 months from completion of parent protocol EOS Visit
  Time from first injection to eGFR <15 mL/min/1.73m² using the 2009 CKD-EPI serum creatinine equation.
Time from first injection to chronic dialysis. | 60 months from completion of parent protocol EOS Visit
  Time from first injection to chronic dialysis
Time from first injection to renal transplant | 60 months from completion of parent protocol EOS Visit
  Time from first injection to renal transplant
Time from first injection to a cardiovascular death. | 60 months from completion of parent protocol EOS Visit
  Time from first injection to a cardiovascular death.
Time from first injection to a renal death. | 60 months from completion of parent protocol EOS Visit
  Time from first injection to a renal death.
Percent of participants who have the same or reduced 5-year risk of end stage renal disease (ESRD) at Months 12, 24, 36, 48, and 60. | 60 months from completion of parent protocol EOS Visit
  Percent of participants who have the same or reduced 5-year risk of end stage renal
Percent of participants who have the same or reduced 2-year risk of end stage renal disease at Months 12, 24, 36, 48, and 60. | 60 months from completion of parent protocol EOS Visit
  Percent of participants who have the same or reduced 2-year risk of end stage renal

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Prokidney
Locations (1):
- Boise Kidney & Hypertension Institute, Meridian, Idaho, United States